CLINICAL TRIAL: NCT00183898
Title: Phase II Study of Oxaliplatin and Xeloda and Cetuximab as First Line Treatment for Metastatic or Unresectable Gastric or Gastroesophageal Junction Cancer
Brief Title: Study of Oxaliplatin and Xeloda and Cetuximab as First Line Treatment for Metastatic or Unresectable Gastric or Gastroesophageal Junction Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: Sanofi (Industry); Roche Global Development (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3G-03-4
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer; Esophageal Cancer
Keywords: Gastroesophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxaliplatin and Capecitabine (Experimental): Oxaliplatin given every 21 days Capecitabine given daily x 14 days every 21 days
  Interventions: Drug: oxaliplatin, capecitabine

INTERVENTIONS:
Drug: oxaliplatin, capecitabine — cetuximab 400 mg/m2, followed by weekly cetuximab 250 mg/m2 with oxaliplatin 130 mg/m2 on day 1 (every 3 weeks) with capecitabine 850 mg/m2 bid, daily on days 1-14, every 3 weeks.

SUMMARY:
This study is for people with advanced gastric or gastroesophageal cancer. This study is being done to find out how long it takes tumors to grow after patients take the drugs capecitabine, oxaliplatin and cetuximab. Capecitabine (also called Xeloda) is a drug that has been approved by the Food and Drug Administration (FDA). Capecitabine has been approved for treatment of cancer of the colon and rectum. Oxaliplatin is another drug approved by the FDA. Oxaliplatin is also approved for treatment of cancer of the colon and rectum. Cetuximab is also a drug approved by the FDA for the treatment of cancer of the colon and rectum, as well as cancer of the head and neck. Capecitabine, oxaliplatin and cetuximab are not approved for gastric or gastroesophageal cancer. They are considered experimental drugs for this study. The purpose of this study is to see how long it takes patients' tumors to progress when they are taking oxaliplatin and capecitabine. Another purpose is to see how many tumors respond to this drug combination. The investigators also want to see how long people live when taking these drugs. The side effects of this drug combination will also be evaluated. This study will also measure the levels of certain genes (the cell's blueprint) in tumors. These genes affect how peoples' bodies react to the cancer drugs. Genes will also be measured in the blood. The investigators want to see how these genes can predict response to these study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced or metastatic gastric or gastroesophageal cancer. Histology must be consistent with adenocarcinoma.
* No previous chemotherapy for metastatic or unresectable disease. Prior adjuvant therapy is allowed, as long as it was completed within six months of study initiation.
* Ability to understand and willingness to sign a written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* SWOG performance status of less than or equal to 2.
* At least one measurable lesion, according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, which has not been irradiated (i.e. newly arising lesions in previously irradiated areas are accepted). Ascites, pleural effusion, and bone metastases are not considered measurable. Minimum indicator lesion size: > 10 mm measured by spiral computed tomography (CT) or > 20 mm measured by conventional techniques.
* Have a negative serum or urine pregnancy test within 7 days prior to initiation of chemotherapy (female patients of childbearing potential).
* Availability of tumor biopsy (paraffin embedded or fresh frozen) at the time of diagnosis and/or prior to study entry is required.
* Patients must agree to use an effective form of birth control while on study and to continue this contraceptive method for 30 days from the date of the last study drug administration.

Exclusion Criteria:

* Pregnant or lactating women.
* Life expectancy of < 3 months.
* Serious, uncontrolled, concurrent infection(s) or illness(es).
* Any prior oxaliplatin treatment.
* Prior unanticipated severe reaction to fluoropyrimidine therapy, known hypersensitivity to 5-fluorouracil or known DPD deficiency.
* Prior unanticipated severe reaction or hypersensitivity to platinum based compounds.
* Completion of previous chemotherapy regimen < four weeks prior to the start of study treatment (within six weeks of study treatment for mitomycin C and nitroureas), or with related toxicities unresolved prior to the start of study treatment.
* Treatment for other carcinomas within the last five years, except for cured non-melanoma skin cancer and treated in-situ cervical cancer.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
* History of clinically significant interstitial lung disease and/or pulmonary fibrosis.
* History of persistent neurosensory disorder including but not limited to peripheral neuropathy
* Evidence of central nervous system (CNS) metastases (unless CNS metastases have been stable for > 3 months) or history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation.
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
* Any of the following laboratory values:

  * Abnormal hematologic values (neutrophils < 1.5 x 10^9/L, platelet count < 100 x 109/L)
  * Impaired renal function (estimated creatinine clearance < 30 ml/min as calculated with Cockroft-Gault equation and serum creatinine > 1.5 x upper normal limit).
  * Serum bilirubin > 1.5 x upper normal limit.
  * ALT, AST > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases).
  * Alkaline phosphatase > 2.5 x upper normal limit (or > 5 x upper normal limit in the case of liver metastases or > 10 x upper normal limit in the case of bone disease).
* Unwillingness to participate or inability to comply with the protocol for the duration of the study.
* Known, existing uncontrolled coagulopathy
* Prior therapy which specifically and directly targets the EGFR pathway.
* Prior severe infusion reaction to a monoclonal antibody

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-12-28 (Actual); Primary Completion 2013-02-04 (Actual); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of patients, with advanced gastric or gastroesophageal junction cancer treated with a combination of capecitabine and oxaliplatin, that have progressive disease within four months of the start of treatment | every 2 cyclec

SECONDARY OUTCOMES:
To determine the time to progression, overall response rate and overall survival in patients with advanced gastric or gastroesophageal junction cancer treated with a combination of capecitabine and oxaliplatin | every 2 cycles
To assess the toxicity of this regimen | every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C./Norris Comprehensive Cancer Center
Locations (1):
- U.S.C./Norris Comprehensive Cancer Center, Los Angeles, California, United States